CLINICAL TRIAL: NCT02384941
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of LX4211 as Adjunct Therapy in Adult Patients With Type 1 Diabetes Mellitus Who Have Inadequate Glycemic Control With Insulin Therapy
Brief Title: Efficacy, Safety, and Tolerability Study of Sotagliflozin as Adjunct Therapy in Adult Patients With Type 1 Diabetes Mellitus Who Have Inadequate Glycemic Control With Insulin Therapy
Acronym: inTandem1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LX4211.1-309-T1DM
Record Dates: First submitted 2015-02-23; First posted 2015-03-10 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Two placebo-matching sotagliflozin tables, orally for 24 weeks followed by a 28 week extension period.
  Interventions: Drug: Placebo
- Sotagliflozin 200 milligrams (mg) (Experimental): Sotagliflozin 200 mg (one 200 mg tablet and one placebo tablet), orally, for 24 weeks followed by a 28 week extension period.
  Interventions: Drug: Placebo; Drug: Sotagliflozin
- Sotagliflozin 400 mg (Experimental): Sotagliflozin 400 mg (two 200 mg tablets), orally, for 24 weeks followed by a 28 week extension period.
  Interventions: Drug: Sotagliflozin

INTERVENTIONS:
Drug: Placebo — Placebo once daily, before first meal of the day.
  Arms: Placebo; Sotagliflozin 200 milligrams (mg)
Drug: Sotagliflozin — Sotagliflozin once daily, before first meal of the day.
  Other Names: LX4211
  Arms: Sotagliflozin 200 milligrams (mg); Sotagliflozin 400 mg

SUMMARY:
This Phase 3 study was intended to demonstrate superiority of either sotagliflozin high dose or low dose versus placebo on glycosylated hemoglobin A1C (A1C) reduction at Week 24 when used as an adjunct in adult participants with type 1 diabetes mellitus (T1D) who have inadequate glycemic control with insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants had given written informed consent to participate in the study in accordance with local regulations.
* Adult participants 18 years and older with a diagnosis of T1D made at least 1 year prior to informed consent.
* Participants were being treated with insulin or insulin analog delivered. via continuous subcutaneous insulin infusion (CSII) or multiple daily injections (MDI).
* Willing and able to perform self-monitored blood glucose (SMBG) and complete the study diary as required per protocol.
* At the Screening Visit, A1C must be between 7.0% to 11.0%.
* Females of childbearing potential must use an adequate method of contraception and have a negative pregnancy test .

Exclusion Criteria:

* Use of antidiabetic agent other than insulin or insulin analog at the time of screening.
* Use of sodium-glucose cotransporter (SGLT) inhibitors within 8 weeks prior to randomization.
* Chronic systemic corticosteroid use.
* Type 2 diabetes mellitus (T2D), or severely uncontrolled T1D as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 793 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sawhney, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (70):
- United States (58):
  - Lexicon Investigational Site, Birmingham, Alabama
  - Lexicon Investigational Site, Little Rock, Arkansas
  - Lexicon Investigational Site, Escondido, California
  - Lexicon Investigational Site, Greenbrae, California
  - Lexicon Investigational Site, Huntington Beach, California
  - Lexicon Investigational Site, La Jolla, California
  - Lexicon Investigational Site, Los Angeles, California
  - Lexicon Investigational Site, Orange, California
  - Lexicon Investigational Site, Palm Springs, California
  - Lexicon Investigational Site, San Mateo, California
  - Lexicon Investigational Site, Tarzana, California
  - Lexicon Investigational Site, Tustin, California
  - Lexicon Investigational Site, Walnut Creek, California
  - Lexicon Investigational Site, Aurora, Colorado
  - Lexicon Investigational Site, Longmont, Colorado
  - Lexicon Investigational Site, Fleming Island, Florida
  - Lexicon Investigational Site, Jacksonville, Florida
  - Lexicon Investigational Site, New Port Richey, Florida
  - Lexicon Investigational Site, Ormond Beach, Florida
  - Lexicon Investigational Site, West Palm Beach, Florida
  - Lexicon Investigational Site, Atlanta, Georgia
  - Lexicon Investigational Site, Lawrenceville, Georgia
  - Lexicon Investigational Site, Roswell, Georgia
  - Lexicon Investigational Site, Honolulu, Hawaii
  - Lexicon Investigational Site, Crystal Lake, Illinois
  - Lexicon Investigational Site, Elgin, Illinois
  - Lexicon Investigational Site, Springfield, Illinois
  - Lexicon Investigational Site, Topeka, Kansas
  - Lexicon Investigational Site, Lexington, Kentucky
  - Lexicon Investigational Site, Bangor, Maine
  - Lexicon Investigational Site, Baltimore, Maryland
  - Lexicon Investigational Site, Boston, Massachusetts
  - Lexicon Investigational Site, Detroit, Michigan
  - Lexicon Investigational Site, Chesterfield, Missouri
  - Lexicon Investigational Site, St Louis, Missouri
  - Lexicon Investigational Site, Omaha, Nebraska
  - Lexicon Investigational Site, Henderson, Nevada
  - Lexicon Investigational Site, Las Vegas, Nevada
  - Lexicon Investigational Site, Albany, New York
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Asheville, North Carolina
  - Lexicon Investigational Site, Chapel Hill, North Carolina
  - Lexicon Investigational Site, Morehead City, North Carolina
  - Lexicon Investigational Site, Columbus, Ohio
  - Lexicon Investigational Site, Oklahoma City, Oklahoma
  - Lexicon Investigational Site, Portland, Oregon
  - Lexicon Investigational Site, Greer, South Carolina
  - Lexicon Investigational Site, Rapid City, South Dakota
  - Lexicon Investigational Site, Chattanooga, Tennessee
  - Lexicon Investigational Site, Memphis, Tennessee
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, Dallas, Texas
  - Lexicon Investigational Site, Houston, Texas
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Schertz, Texas
  - Lexicon Investigational Site, Chesapeake, Virginia
  - Lexicon Investigational Site, Renton, Washington
  - Lexicon Investigational Site, Seattle, Washington
- Canada (12):
  - Lexicon Investigational Site, Calgary, Alberta
  - Lexicon Investigational Site, Vancouver, British Columbia
  - Lexicon Investigational Site, Winnipeg, Manitoba
  - Lexicon Investigational Site, Halifax, Nova Scotia
  - Lexicon Investigational Site, Barrie, Ontario
  - Lexicon Investigational Site, Hamilton, Ontario
  - Lexicon Investigational Site, London, Ontario
  - Lexicon Investigational Site, Ottawa, Ontario
  - Lexicon Investigational Site, Thornhill, Ontario
  - Lexicon Investigational Site, Toronto, Ontario
  - Lexicon Investigational Site, Montreal, Quebec
  - Lexicon Investigational Site, Saint-Laurent, Quebec

REFERENCES:
- [Derived] Peters AL, McGuire DK, Danne T, Kushner JA, Rodbard HW, Dhatariya K, Sawhney S, Banks P, Jiang W, Davies MJ, Lapuerta P. Diabetic Ketoacidosis and Related Events With Sotagliflozin Added to Insulin in Adults With Type 1 Diabetes: A Pooled Analysis of the inTandem 1 and 2 Studies. Diabetes Care. 2020 Nov;43(11):2713-2720. doi: 10.2337/dc20-0924. Epub 2020 Sep 14. PMID 32928957
- [Derived] Danne T, Joish VN, Afonso M, Banks P, Sawhney S, Lapuerta P, Davies MJ, Buse JB, Lin D, Reaney M, Guillonneau S, Snoek FJ, Bailey TS, Polonsky WH. Improvement in Patient-Reported Outcomes in Adults with Type 1 Diabetes Treated with Sotagliflozin plus Insulin Versus Insulin Alone. Diabetes Technol Ther. 2021 Jan;23(1):70-77. doi: 10.1089/dia.2020.0068. PMID 32721228
- [Derived] Ervin C, Joish VN, Evans E, DiBenedetti D, Reaney M, Preblick R, Castro R, Danne T, Buse JB, Lapuerta P. Insights Into Patients' Experience With Type 1 Diabetes: Exit Interviews From Phase III Studies of Sotagliflozin. Clin Ther. 2019 Nov;41(11):2219-2230.e6. doi: 10.1016/j.clinthera.2019.09.003. Epub 2019 Oct 3. PMID 31587812
- [Derived] Danne T, Cariou B, Buse JB, Garg SK, Rosenstock J, Banks P, Kushner JA, McGuire DK, Peters AL, Sawhney S, Strumph P. Improved Time in Range and Glycemic Variability With Sotagliflozin in Combination With Insulin in Adults With Type 1 Diabetes: A Pooled Analysis of 24-Week Continuous Glucose Monitoring Data From the inTandem Program. Diabetes Care. 2019 May;42(5):919-930. doi: 10.2337/dc18-2149. Epub 2019 Mar 4. PMID 30833371
- [Derived] Buse JB, Garg SK, Rosenstock J, Bailey TS, Banks P, Bode BW, Danne T, Kushner JA, Lane WS, Lapuerta P, McGuire DK, Peters AL, Reed J, Sawhney S, Strumph P. Sotagliflozin in Combination With Optimized Insulin Therapy in Adults With Type 1 Diabetes: The North American inTandem1 Study. Diabetes Care. 2018 Sep;41(9):1970-1980. doi: 10.2337/dc18-0343. Epub 2018 Jun 24. PMID 29937430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 75 study sites in 2 countries from March 2015 to February 2017.
Pre-assignment Details: 1099 participants were screened and 793 participants with Type 1 diabetes mellitus who had inadequate glycemic control with insulin therapy were randomized into three treatment groups: Placebo, Sotagliflozin 200 mg, Sotagliflozin 400 mg.
Groups:
- Placebo: Two placebo-matching sotagliflozin tablets, once daily, orally for 24 weeks followed by a 28 week extension period.
- Sotagliflozin 200 mg: Sotagliflozin 200 mg (one 200 mg tablet and one placebo tablet), once daily, orally, for 24 weeks followed by a 28 week extension period.
- Sotagliflozin 400 mg: Sotagliflozin 400 mg (two 200 mg tablets), once daily, orally, for 24 weeks followed by a 28 week extension period.
Period: Overall Study
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Started | 268 | 263 | 262
Completed | 218 | 228 | 221
Not Completed | 50 | 35 | 41
Not completed — Adverse Event | 11 | 13 | 17
Not completed — Lost to Follow-up | 3 | 2 | 1
Not completed — Non-Compliance With Study Drug | 2 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 19 | 20
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Other than specified above | 4 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent to treat (mITT) analysis set included all randomly assigned participants who have taken at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg | Total
Number analyzed (Participants) | 268 | 263 | 262 | 793
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.72) | 46.6 (13.48) | 46.4 (13.12) | 46.1 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 137 | 142 | 410
  Male | 137 | 126 | 120 | 383
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 4 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 0 | 4
  Black or African American | 9 | 11 | 8 | 28
  White | 244 | 241 | 246 | 731
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 6 | 19
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: percentage of A1C] | 7.54 (0.712) | 7.61 (0.735) | 7.56 (0.724) | 7.57 (0.723)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 87.30 (17.709) | 86.96 (18.539) | 86.50 (18.004) | 86.92 (18.065)
Baseline Daily Total Insulin Dose [Mean (Standard Deviation); unit: International Unit per kilogram (IU/kg)] | 0.74 (0.357) | 0.72 (0.386) | 0.72 (0.335) | 0.73 (0.360)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] | 29.55 (5.188) | 29.81 (5.686) | 29.63 (5.297) | 29.66 (5.387)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 24.2 (12.38) | 25.0 (13.15) | 24.0 (12.88) | 24.4 (12.80)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. Least square (LS) means were obtained from a mixed-effects model for repeated measures (MMRM) that included fixed, categorical effects of treatment, randomization strata of insulin delivery method (MDI, CSII), randomization strata of Week -2 A1C (<= 8.5%, >8.5%), time (study week), a treatment-by-time interaction, and baseline A1C-by-time interaction as a covariate. A negative change from Baseline (a lower A1C value at Week 24) indicates an improvement.
Time Frame: Baseline to Week 24
Population: Modified intent to treat (mITT) analysis set included all randomly assigned participants who have taken at least 1 dose of study drug. Here, "Overall Number of Participants" Analyzed signified participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of A1C
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 246 | 245 | 242
percentage of A1C | -0.07 (0.036) | -0.43 (0.036) | -0.48 (0.036)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.36, Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.41, Standard Error of Mean 0.047

2. Secondary Outcome: Percentage of Participants With A1C <7.0% (at Week 24) and No Episode of Severe Hypoglycemia and No Episode of Diabetic Ketoacidosis (DKA) Upto Week 24
Description: Blood samples were collected for the assessment of Hemoglobin A1C to determine the participants with A1C value <7.0%. A central blinded adjudication process determined whether participants experienced either DKA or Severe Hypoglycemia. Only positively adjudicated severe hypoglycemia and diabetic ketoacidosis were included in the analysis.
Time Frame: Baseline to Week 24
Population: Analysis performed on mITT analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 268 | 263 | 262
percentage of participants | 21.6 | 33.5 | 43.5
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints were reported. The hierarchical testing sequence continued only when previous endpoint of each treatment comparison was statistically significant at 0.05 level; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Threshold for significance < 0.05; Percentage difference = 11.8, 95% CI 2-sided [4.28 to 19.36]
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant for the relevant compared arms); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Threshold for significance < 0.05; Percentage difference = 21.9, 95% CI 2-sided [14.10 to 29.64]

3. Secondary Outcome: Absolute Change From Baseline in Body Weight at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model. A negative change from Baseline indicates a loss in body weight from Baseline to Week 24.
Time Frame: Baseline to Week 24
Population: Analysis performed on mITT analysis set. Here, "Overall Number of Participants Analyzed" signified participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 244 | 245 | 242
kilograms (kg) | 0.78 (0.187) | -1.57 (0.188) | -2.67 (0.188)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -2.35, 95% CI 2-sided [-2.85 to -1.85], Standard Error of Mean 0.256
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -3.45, 95% CI 2-sided [-3.95 to -2.94], Standard Error of Mean 0.256

4. Secondary Outcome: Change From Baseline in Mean Daily Bolus Insulin Dose at Week 24
Description: The mean bolus insulin dose in international units per day (IU/day) for Week 24 was the average over the 3 to 5 days prior to the Week 24 visit. The Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post Baseline values. A negative change from Baseline indicated a reduction in the amount of bolus insulin used between Baseline and Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: IU/day
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 241 | 242 | 242
IU/day | -0.84 (0.688) | -2.33 (0.692) | -4.13 (0.692)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 200 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.10, MMRM — Threshold for significance < 0.05; Least squares mean difference = -1.50, 95% CI 2-sided [-3.30 to 0.30], Standard Error of Mean 0.917
Statistical Analysis 2: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -3.30, 95% CI 2-sided [-5.09 to -1.50], Standard Error of Mean 0.916

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: The Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model including all available post baseline values. A negative change from baseline indicates a lower glucose at Week 24 compared to baseline.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Groups:
- Placebo: Two placebo-matching sotagliflozin tables, once daily, orally for 24 weeks followed by a 28 week extension period.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 245 | 245 | 242
millimole per liter (mmol/L) | 0.21 (0.191) | -0.34 (0.192) | -0.78 (0.193)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.99, 95% CI 2-sided [-1.50 to -0.48], Standard Error of Mean 0.260

6. Secondary Outcome: Change From Baseline in Diabetes Total Treatment Satisfaction Scores as Measured by Total Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) Scores at Week 24
Description: DTSQs is a diabetes-specific measure used to evaluate overall treatment satisfaction and perception of hyperglycemia and hypoglycemia events. It consists of 8 items and the response categories for all items were on a 7-point likert scale.The DTSQs response options ranged from 0 (very dissatisfied) to 6 (very satisfied). Responses to item 1, 4, 5, 6, 7 and 8 were summarized to determine the total treatment satisfaction score which ranged from 0 (very dissatisfied) to 36 (very satisfied), with a higher score corresponding to higher satisfaction . LS means were obtained from MMRM model including all available post baseline values. A positive change from baseline indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 237 | 240 | 233
units on a scale | -0.4 (0.30) | 2.1 (0.31) | 2.1 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = 2.5, 95% CI 2-sided [1.8 to 3.3], Standard Error of Mean 0.40

7. Secondary Outcome: Change From Baseline in Diabetes Distress Scores as Measured by 2-item Diabetes Distress Screening Scale (DDS2) Scores at Week 24
Description: The DDS2 is a 2-item diabetes distress screening instrument where respondents rated, on a 6-point scale, the degree to which the following items caused distress: (1) feeling overwhelmed by the demands of living with diabetes, and (2) feeling that I am often failing with my diabetes regimen using a 6-point scale: where 1=no distress to 6=severe distress for a total possible score of 2 (not a problem) to 12 (very serious problem), with higher score corresponding to higher distress. LS means were obtained from MMRM model including all available post baseline values. A negative change from baseline indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 243 | 244 | 242
units on a scale | 0.3 (0.11) | -0.4 (0.11) | -0.5 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Sotagliflozin 400 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — Threshold for significance < 0.05; Least squares mean difference = -0.8, 95% CI 2-sided [-1.0 to -0.5], Standard Error of Mean 0.14

8. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 24
Description: Baseline value was defined as the last value collected prior to the first dose of double-blind study medication. LS means were obtained from MMRM model. A negative percent change from baseline indicates a loss in body weight from baseline to Week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
Number analyzed (Participants) | 244 | 245 | 242
percent change | 0.92 (0.212) | -1.87 (0.213) | -3.10 (0.213)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) to 30 days after end of treatment or end of follow up (Up to 53 Weeks)
Description: Analysis performed on safety population which includes participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Sotagliflozin 200 mg | Sotagliflozin 400 mg
All-Cause Mortality (participants affected / at risk) | 1/268 | 0/263 | 0/262
Serious Adverse Events (participants affected / at risk) | 20/268 | 27/263 | 29/262
Other Adverse Events (participants affected / at risk) | 129/268 | 132/263 | 130/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=268) | Sotagliflozin 200 mg (N=263) | Sotagliflozin 400 mg (N=262)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acetonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 12 (13) | 14 (14)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (7) | 3 (5) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Foot amputation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=268) | Sotagliflozin 200 mg (N=263) | Sotagliflozin 400 mg (N=262)
Blood ketone body increased (Investigations) | 2 (2) | 10 (20) | 14 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 6 (6) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 19 (21) | 22 (26) | 29 (41)
Nausea (Gastrointestinal disorders) | 18 (21) | 17 (23) | 18 (24)
Sinusitis (Infections and infestations) | 13 (16) | 14 (20) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 43 (52) | 33 (38) | 33 (46)
Urinary tract infection (Infections and infestations) | 18 (23) | 25 (34) | 9 (14)
Viral upper respiratory tract infection (Infections and infestations) | 29 (33) | 34 (41) | 24 (29)
Vulvovaginal mycotic infection (Infections and infestations) | 6 (8) | 13 (18) | 21 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.